CLINICAL TRIAL: NCT07206758
Title: A Phase I Study Evaluating the Safety, Efficacy, Pharmacokinetics and Pharmacokinetics of SHR-2173 Injection in Patients With Primary Immune Thrombocytopenia
Brief Title: Phase I Study of SHR-2173 Injection in Patients With Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2173-105
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-2173 Injection (Experimental)
  Interventions: Drug: SHR-2173 Injection

INTERVENTIONS:
Drug: SHR-2173 Injection — SHR-2173 injection treatment

SUMMARY:
Evaluate the safety and tolerance of multiple subcutaneous injections of SHR-2173 in ITP patients

ELIGIBILITY:
Inclusion Criteria:

1. Participants must fully understand the trial content, procedures, and potential adverse reactions, and voluntarily sign a written informed consent form (ICF).
2. Age at signing the ICF must be ≥ 18 years (including the boundary value), regardless of gender.
3. Confirmed diagnosis of primary ITP for at least 3 months at screening.
4. Previous treatment with corticosteroids.
5. At the last ITP treatment, participants experienced loss of remission, no remission, relapse after remission, or intolerance.
6. Platelet count <30×10⁹/L at screening with clinical assessment indicating treatment necessity
7. Participants must have adequate organ function
8. Clinically stable condition with World Health Organization (WHO) bleeding scale grade 0-1
9. Female participants of childbearing potential or male participants with fertile partners must refrain from sperm/ova donation from ICF signing until 12 weeks after last dose and agree to protocol-specified contraceptive measures

Exclusion Criteria:

1. Diagnosis of secondary thrombocytopenia or concomitant autoimmune hemolytic anemia
2. Received platelet transfusion, whole blood transfusion, plasma exchange, or any other emergency treatment drugs within 14 days prior to the first infusion of SHR-2173
3. Received immunosuppressants (other than corticosteroids) such as Janus kinase [JAK] inhibitors or Bruton tyrosine kinase [BTK] inhibitors within either 5 times the drug elimination half-life or 14 days prior to the first infusion of SHR-2173 (whichever is longer)
4. Previous treatment with SHR-2173
5. Screening prothrombin time or activated partial thromboplastin time outside the normal range; concurrent coagulation disorders and/or receiving antiplatelet or anticoagulant medications (e.g., warfarin, clopidogrel, novel oral anticoagulants), except for low-dose acetylsalicylic acid
6. History of any thrombotic or embolic events within 12 months prior to the first administration, or clinical symptoms and history suggesting thrombophilia
7. Current life-threatening bleeding (related to thrombocytopenia) or expected to require emergency treatment within one week after randomization
8. Active viral, bacterial, or other infections (including tuberculosis [TB]) requiring systemic treatment at screening, or SARS-CoV-2 infection during screening, or history of clinically significant recurrent infections
9. Received live or attenuated live vaccines within 8 weeks prior to the first administration of SHR-2173, or planned to receive live/attenuated vaccinations during the trial
10. Received live or attenuated live vaccines within 8 weeks prior to the first administration of SHR-2173, or planned to receive live/attenuated vaccinations during the trial
11. Diagnosis of myelodysplastic syndrome; history of or current malignancy within 5 years prior to screening (except for cured non-melanoma skin cancer, in situ carcinoma [e.g., cervical, breast, bladder, prostate cancer], and cancers in complete remission for at least 5 years with no evidence of recurrence)
12. Previous splenectomy
13. Previous allogeneic stem cell or organ transplantation (except for corneal transplantation ≥ 3 months prior to screening); known or suspected history of immunosuppression
14. Planned surgery during the dosing period
15. Any severe and/or unstable pre-existing medical, psychiatric, or other conditions that the investigator judges may interfere with patient safety, obtaining informed consent, or compliance with study procedures
16. Allergic constitution (e.g., allergies to two or more drugs, foods, or pollens) or known hypersensitivity (immediate or delayed) or atopic reactions to the study drug (including excipients, monoclonal antibodies)
17. Concurrent participation in other investigational studies within either 30 days prior to enrollment or 5 half-lives of the investigational drug (whichever is longer)
18. Females who are lactating or pregnant (positive serum or urine β-human chorionic gonadotropin [hCG]) at screening or on Day 1 of Week 1 prior to administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) and adverse events of special concern (AESI) | About in the ninth month
The severity of adverse events (AE) and serious adverse events (SAE) and adverse events of special concern (AESI) | About in the ninth month
Changes in abnormal indicators in laboratory inspection | About in the ninth month

SECONDARY OUTCOMES:
Percentage of subjects achieving remission response at week 13 of the treatment period | About in the fourth month
Percentage of subjects achieving remission response at week 25 of the treatment period | About in the sixth month
Percentage of participants achieving remission response at any time during the treatment period | About in the ninth month
Proportion of participants achieving confirmed remission after SHR-2173 injection treatment | About in the ninth month
Time from first SHR-2173 injection treatment to confirmed remission | About in the ninth month
Duration from first confirmed remission to date of remission loss | About in the ninth month
Number and severity of bleeding events | About in the ninth month
Percentage of participants requiring rescue therapy | About in the ninth month
Serum concentration of SHR-2173 | About in the ninth month
Anti-SHR-2173 antibodies | About in the ninth month
Serum immunoglobulin levels | About in the ninth month
Count and percentage of B cells and subsets in peripheral blood | About in the ninth month

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided